CLINICAL TRIAL: NCT04765397
Title: The Effect of Bipolar and Monopolar Resectoscope Use on Optic Nerve Diameter in Transurethral Resection Procedures Under Spinal Anesthesia
Brief Title: Different Resectoscopes Effects to Optic Nerve Sheath Diameter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Umran Karaca, Medical Doctor, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Bursa Yüksek Ihtisas EAH
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Optic Nerve Sheath Diameter
Keywords: Monopolar Resectoscope; Bipolar Resectoscope

STUDY DESIGN:
Intervention Model Description: According to the resectoscopes used during the operation, patients will be divided into 2 groups as Monopolar one (Group M) and Bipolar one (Group B).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group M (Active Comparator): Patients are in this group with monopolar technique according to the resectoscope technique used by the surgeon.Demographic data of the patients, mean arterial pressure (MAP), pulse minute number (NDS), peripheral oxygen saturation (SpO2), irrigation and intravenous fluid amounts, operation times, serum electrolytes (Na +, K +) and hemoglobin levels were analyzed and recorded.
  Interventions: Procedure: Effect of different resectoscope fluids on optic nerve diameter measured by ultrasound
- Group B (Active Comparator): Patients are in this group with bipolar technique according to the resectoscope technique used by the surgeon.Demographic data of the patients, mean arterial pressure (MAP), pulse minute number (NDS), peripheral oxygen saturation (SpO2), irrigation and intravenous fluid amounts, operation times, serum electrolytes (Na +, K +) and hemoglobin levels were analyzed and recorded.
  Interventions: Procedure: Effect of different resectoscope fluids on optic nerve diameter measured by ultrasound

INTERVENTIONS:
Procedure: Effect of different resectoscope fluids on optic nerve diameter measured by ultrasound — During the operation Blood pressure, pulse minute the number of irrigation solutions used, and intravenous serum amounts, operation time will be saved. If there is an abnormal parameters or increased optic nerve sheath surgical team will be informed.

SUMMARY:
In this study, in patients with benign prostatic hypertrophy, monopolar and transurethral prostate using bipolar techniques in resection; serum electrolytes in the perioperative period, osmolarity can occur in hemodynamic parameters the effect of changes on optic nerve diameter by ultrasonography.

DETAILED DESCRIPTION:
This study is for TURP operation for Benign Prostate Hypertrophy patients. When patient comes to the operating room, routine preparations will be made. Haemodynamic parameters and over-the-eye with Optic nerve diameter will be checked with ultrasound before and 10 minutes after spinal anesthesia. Monopolar for patients according to the preference of the surgical team resectoscope technique or bipolar resectoscope technique will be applied. During the operation Blood pressure, pulse minute the number of irrigation solutions used and the amount of intravenously administered serum, operation time will be saved. Optic nerve sheath diameter after the operation would be checked again. intraoperative and postoperative complications in the waking room (respiratory distress, hypotension, hypertension, bradycardia, tachycardia, vomiting, headache, restlessness, seizure, arrhythmia, vision disorder) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Ages 50-80
* ASA I-II
* Planned TUR-P operation

Exclusion Criteria:

* Heart or respiratory failure
* Koagülation diathesis
* Eyedisease related patients

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
optic nerve sheath diameter(mm) | operation time 3 hours
  A linear 10-5 MHz ultrasound probe (GE Healthcare Logiqe Series) was held on the upper eyelid over the gel carefully. Part of the optical nerve that enters the orbital globe was monitorized in the 2D mode without exerting much pressure. Diameter of the optic nerve sheath was measured 3 mm behind the optic disk using an electronic caliper after the right contrast was found between the retrobulber echogenic fatty tissue and the vertical hypoechogenic band

CONTACTS AND LOCATIONS:
Overall Officials: Ümran K Karaca, MD, Principal Investigator — Bursa Yuksek Ihtisas Training and Research Hospital; Tuğba O Onur, MD, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital; Seyda Ö Özgünay, MD, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital; Sermin E Eminoglu, MD, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital; Ayse Neslihan B Balkaya, MD, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital
Locations (1):
- University of Health Sciences Bursa Yüksek İhtisas Training and Research Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No